CLINICAL TRIAL: NCT05042128
Title: A Randomised, Double-blinded Phase II Study of Gemcitabine and Nab-Paclitaxel With LSTA1 (Certepetide) or Placebo in Patients With Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: The ASCEND Study: Gemcitabine and Nab-Paclitaxel With LSTA1 (Certepetide) or Placebo in Patients With Untreated Metastatic Pancreatic Ductal Adenocarcinoma
Acronym: ASCEND
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Australasian Gastro-Intestinal Trials Group (Network)
Collaborators: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTC0304
Record Dates: First submitted 2021-08-25; First posted 2021-09-13 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A: Standard Care + LSTA1 (1 dose) (Experimental): Participants will receive nab-paclitaxel 125mg/m2; LSTA1 3.2mg/kg IV; and then Gemcitabine 1000mg/m2, on Day 1, 8 and 15 of each cycle. Each cycle will be 28 days.
  Interventions: Drug: LSTA1; Drug: Gemcitabine Injection; Drug: Nab paclitaxel
- Cohort A: Standard Care + Placebo (Placebo Comparator): Participants will receive nab-paclitaxel 125mg/m2; placebo IV; and then Gemcitabine 1000mg/m2, on Day 1, 8 and 15 of each cycle. Each cycle will be 28 days.
  Interventions: Drug: Gemcitabine Injection; Drug: Nab paclitaxel
- Cohort B: Standard Care +LSTA1 (2 doses) (Experimental): Participants will receive nab-paclitaxel 125mg/m2; LSTA1 3.2mg/kg IV; Gemcitabine 1000mg/m2, and then +~4hrs LSTA1 3.2mg/kg IV on Day 1, 8 and 15 of each cycle. Each cycle will be 28 days.
  Interventions: Drug: LSTA1; Drug: Gemcitabine Injection; Drug: Nab paclitaxel
- Cohort B: Standard Care + Placebo (Placebo Comparator): Participants will receive nab-paclitaxel 125mg/m2; placebo IV; Gemcitabine 1000mg/m2, and then +~4hrs matching placebo IV on Day 1, 8 and 15 of each cycle. Each cycle will be 28 days.
  Interventions: Drug: Gemcitabine Injection; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: LSTA1 — LSTA1 is a novel cyclic tumour-penetrating peptide iRGD (internalizing Arginylglycylaspartic acid) which may overcome poor drug delivery by activation of a complex trans-tissue transport pathway, providing an opportunity to overcome this mechanism of resistance in PDAC
  Other Names: CEND-1, certepetide
  Arms: Cohort A: Standard Care + LSTA1 (1 dose); Cohort B: Standard Care +LSTA1 (2 doses)
Drug: Gemcitabine Injection — Chemotherapy drug provided as solution to be administered via IV infusion.
  Other Names: Gemzar
Drug: Nab paclitaxel — Chemotherapy drug provided as solution to be administered via IV infusion.
  Other Names: Abraxane

SUMMARY:
The purpose of the ASCEND clinical trial is to measure the effect of adding LSTA1 (certepetide), compared to placebo, to chemotherapy (gemcitabine and nab-paclitaxel) in patients who have untreated metastatic pancreatic cancer. The study will assess the duration which the cancer remained stable or improved, the number of patients who responded to treatment, overall survival, side effects and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older with histologically confirmed metastatic pancreatic ductal adenocarcinoma or poorly differentiated carcinoma.
* Measurable disease according to RECIST 1.1.
* Archival tumour tissue for tertiary correlative studies (biopsy or resection of primary or metastasis). Fine needle aspirate (FNA) or brushings will not be accepted.
* ECOG performance of 0-1 (Appendix 2)
* Adequate renal and haematological function
* Adequate hepatic function, defined as:

Bilirubin <1.5 X ULN (Upper Limit of Normal), AST or ALT ≤ 5x ULN. If a person was recently stented with improving bilirubin, the person can be randomised with bilirubin up to 3 x ULN provided chemotherapy is not administered until within the stated thresholds.

* Willing and able to comply with all study requirements, including treatment, timing and/or nature of required assessments.
* Study treatment both planned and able to start within 7 days after randomisation
* Signed, written informed consent.

Exclusion Criteria:

* Uncontrolled metastatic disease to the central nervous system. To be eligible, known CNS metastases should have been treated with surgery and/or radiotherapy and the patient should have been receiving a stable dose of steroids for at least 2 weeks prior to randomisation, with no deterioration in neurological symptoms during this time.
* Prior chemotherapy or investigational anti-cancer therapy for metastatic pancreatic adenocarcinoma. Prior treatments with curative intent or for locally advanced disease are allowed, provided the last dose of chemotherapy was administered more than 6 months prior to randomisation.
* Prior radiotherapy or major surgery (as defined by local investigator) within 14 days of starting treatment.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anti-cancer therapy with the exception of alopecia, vitiligo and the laboratory values defined in the inclusion criteria. Participants with Grade ≥2 peripheral neuropathy are not allowed.
* Concurrent use of any other anti-cancer therapy including chemotherapy, targeted therapy, immunotherapy or biological agents.
* Known allergy or hypersensitivity to any of the study drugs and excipients.
* Any significant active infection, including chronic active hepatitis B, hepatitis C, or HIV. Participants with known Hepatitis B/C infection will be allowed to participate providing evidence of viral suppression has been documented and the patient remains on appropriate anti-viral therapy.
* History of prior or synchronous malignancy within 2 years prior to randomisation, except:

  1. Malignancy that was treated with curative intent and for which there has been no known active disease for ≥2 years prior to randomisation.
  2. Curatively treated non-melanoma skin cancer, cervical cancer in situ, superficial transitional cell carcinoma of the bladder, stage 1 endometrial carcinoma, prostatic intraepithelial neoplasia, low-grade papillary thyroid cancer, untreated localised very low risk or low risk prostate cancer under observation.
* Concurrent illness, including severe infection that may jeopardise the ability of the person to undergo the procedures outlined in this protocol with reasonable safety.
* Neuroendocrine pancreatic carcinoma.
* Life expectancy of less than 3 months.
* Pregnancy, lactation, or inadequate contraception. Women must be post-menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to randomisation. Men must use a reliable means of contraception.
* Serious medical or psychiatric conditions that might limit the ability of the person to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of randomization to 18 months later, or death
  Period of time from randomization to the date of first evidence of disease progression, the occurrence of new disease or death from any cause

SECONDARY OUTCOMES:
Overall Survival | From date of randomization to 18 months later, or death
  Period of time from randomization to date of death from any cause, or the date of last known follow-up alive
Objective Tumour Response Rate | From date of randomization to 18 months later, or death
  The number of participants with documented partial or complete response (PR or CR) divided by the number of participants evaluable for response as defined as per the RECIST version 1.1 criteria
Patient-reported Outcomes | Completed at baseline, then every 8 weeks from randomization until and at disease progression (to a maximum of 48 months).
  Completion of the EORTC QLQ-C30 questionnaire. 30 questions; 28 on a 1-4 scale (Higher scores indicative of poorer quality of life), 2 on a 1-7 scale (higher scores indicative of better health/quality of life).
Patient-reported Outcomes | Completed at baseline, then every 8 weeks from randomization until and at disease progression (to a maximum of 48 months).
  Completion of the QLQ-PAN26 questionnaire. 26 questions on a 1-4 scale (Higher scores indicative of poorer quality of life)
Incidence of Treatment-Emergent Adverse Events (Patient Safety) | From date of randomization until 30 days after final treatment visit
  Record of all adverse events (including SAEs) that patients experience

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Dean, Study Chair — St John of God Hospital; Timothy Price, Study Chair — The Queen Elizabeth Hospital
Locations (24):
- Australia (22):
  - Border Medical Oncology, Albury, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Monash Medical Centre, Clayton, New South Wales
  - Lake Macquarie Private Hospital, Gateshead, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Newcastle Private Hospital, Newcastle, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - Icon Cancer Centre Wesley, Auchenflower, Queensland
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Royal Brisbane and Womens Hospital, Herston, Queensland
  - ICON Cancer Centre, Gold Coast University Hospital, Southport, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Queen Elizabeth Hospital, Woodville South, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Northern Health, Epping, Victoria
  - Warringal Private Hospital, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Frankston Hospital, Melbourne, Victoria
  - Epworth Healthcare, Richmond, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God, Subiaco, Western Australia
- New Zealand (2):
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dean A, Gill S, McGregor M, et al. 1528P Phase I trial of the first-in-class agent CEND-1 in combination with gemcitabine and nab-paclitaxel in patients with metastatic pancreatic cancer. Annals of Oncology 2020; 31: S941.